CLINICAL TRIAL: NCT03236207
Title: Hypoallergenicity Evaluation of a New Extensively Hydrolyzed Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16.16.CLI
Record Dates: First submitted 2017-07-19; First posted 2017-08-01 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test infant formula (Experimental): Test non-commercial extensively hydrolyzed infant formula with HMOs
  Interventions: Other: Test extensively hydrolyzed formula
- Control infant formula (Active Comparator): Control non-commercial extensively hydrolyzed infant formula without HMOs
  Interventions: Other: Control extensively hydrolyzed formula

INTERVENTIONS:
Other: Test extensively hydrolyzed formula — extensively hydrolyzed formula with HMOs
  Arms: Test infant formula
Other: Control extensively hydrolyzed formula — extensively hydrolyzed formula without HMOs
  Arms: Control infant formula

SUMMARY:
Infants/children with cow's milk allergy will take part in 2 double-blinded placebo-controlled food challenges (DBPCFC) of 2 extensively hydrolyzed formulas in random order. If both food challenges are passed, subjects will be asked to consume the Test formula in an at-home open challenge for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Born at term (>36 weeks gestation)
* 2 months to <4 years of age at enrollment
* Documented CMA within 6 months prior to enrollment
* Otherwise healthy
* Having obtained his/her legal representative's informed consent

Exclusion Criteria:

* Children consuming mother's milk at the time of inclusion and during the trial
* Any chromosomal or major congenital anomalies
* Chronic medical diseases (ie seizure disorders, chronic lung disease, heart problems (heart murmurs okay))
* Immunodeficiency
* Anaphylaxis to any food
* Receiving free amino acid formula
* Subject who in the Investigator's assessment cannot be expected to adhere to the study protocol
* Currently participating in another clinical trial

Ages: 2 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
allergic reaction post DBPCFC | 2 hours
  subjects will be observed during and for at least 2 hours after the food challenge for any allergic reaction symptoms which will be documented by investigators

SECONDARY OUTCOMES:
stool characteristics | 1 week
  collected on daily diaries
formula intake | 1 week
  amount of formula ingested daily
adverse events | 1 week
  adverse events as reported by caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nowak-Wegrzyn, MD, Principal Investigator — Mt Sinai
Locations (12):
- United States (12):
  - Hoag Medical Group, Huntington Beach, California
  - Stanford University, Mountain View, California
  - Clinical Research Institute, Plymouth, Minnesota
  - Midwest Clinical Research, St Louis, Missouri
  - Breathe America, Albuquerque, New Mexico
  - Northwell Health System, Great Neck, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Carolina ENT, Orangeburg, South Carolina
  - Memphis & Shelby County Pediatrics, Memphis, Tennessee
  - Houston Clinical Research Associates, Houston, Texas
  - Allergy Asthma Research Institute, Waco, Texas

IPD SHARING:
Plan to Share IPD: No